CLINICAL TRIAL: NCT03926234
Title: The Reliability and Validity of a Four-level Chinese Emergency Triage Scale in Mainland China
Brief Title: Effectiveness of a Four-level Chinese Emergency Triage Scale in Mainland China
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Tongji Hospital (Other); Henan Provincial People's Hospital (Other); Second Affiliated Hospital of Chongqing Mecical University (Unknown); First People's Hospital of Hangzhou (Other); Second People's Hospital of Hangzhou (Unknown); Changxing People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018ZH012
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Emergencies; Triage
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- emergency triage patients: triage Level I triage Level II triage Level III triage Level IV
  Interventions: Other: Four-level Chinese Emergency triage scale

INTERVENTIONS:
Other: Four-level Chinese Emergency triage scale — a four-level category system, i.e. life-threatening (Level I), emergent (Level II), urgent (Level III) and semi-urgent (Level IV) . This system contains critical indicators (cardiac arrest, shock, and apnea), high risk indicators (ACS and DKA), single objective indicators (SBP, RR, HR, and SpO2) and MEWS (synthesis indicator). According to patients' health care problems, patients are rated by nurses into one of the four mentioned levels.

SUMMARY:
Inter-rater reliability between experts and triage nurses was assessed in 484 emergency patients. The criterion-related validity was evaluated in other 30687 emergency patients, based on emergency department (ED) mortality, the length of stay in ED, the number of discharge, and hospitalization (intensive care/general ward).

ELIGIBILITY:
Inclusion Criteria:

* Patients, older than 14 years and admitted to the ED, were eligible for this study.

Exclusion Criteria:

* Gynecologic and obstetric emergencies
* Patients, who left against medical advice or hadn't been aided by a doctor

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligibility emergency patients
Sampling Method: Probability Sample
Enrollment: 30687 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability | 2019-10-1
  inter-rater reliability as the agreement between triage nurses and experts
emergency department (ED) mortality | 2019-12-31
the number of discharge | 2019-12-31

SECONDARY OUTCOMES:
the number of hospitalization | 2019-12-31

CONTACTS AND LOCATIONS:
Locations (1):
- SAHZhejiangU, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided